CLINICAL TRIAL: NCT06151522
Title: 90% Effective Dose of Phenylephrine Infusions for Preventing Postspinal Anesthesia Hypotension Under Intensive and Standard Treatment During Cesarean Section
Brief Title: 90% Effective Dose of Phenylephrine Infusions Under Intensive and Standard Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2024-4
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Adverse Effect
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Other): The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Alpha-Agonist
- Intensive group (Other): The maternal systolic blood pressure was consistently maintained above 90% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: α-adrenergic receptor agonist

INTERVENTIONS:
Drug: Alpha-Agonist — An initial infusion dose of prophylactic phenylephrine (0.625 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.125 ug/kg/min of prophylactic phenylephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: norepinephrine
  Arms: Standard group
Drug: α-adrenergic receptor agonist — An initial infusion dose of prophylactic phenylephrine (0.625 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.125 ug/kg/min of prophylactic phenylephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: norepinephrine
  Arms: Intensive group

SUMMARY:
The objective of this study is to investigate the 90% effective dose of phenylephrine infusions for preventing postspinal anesthesia hypotension under intensive and standard treatment during cesarean section

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. The 2016 ASA guidelines for obstetric anesthesia suggest avoiding hypotension following spinal anesthesia in women and emphasize the use of vasopressors, specifically alpha-receptor agonists, as the preferred strategy to prevent and manage post-spinal anesthesia hypotension. The 2018 International Consensus in the United Kingdom and Northern Ireland recommends maintaining maternal systolic blood pressure above 90% of the baseline value following lumbar anesthesia, while avoiding dropping below 80% of the baseline value. Currently, the threshold for maintaining blood pressure above 80% of the baseline value is widely adopted as a standard; however, limited evidence supports the advantage of sustaining maternal blood pressure above 90% of the baseline value. The objective of this study is to investigate the 90% effective dose of phenylephrine infusions for preventing postspinal anesthesia hypotension under intensive and standard treatment during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥180 mmHg
* Hemoglobin < 7g/dl

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ED50 and ED90 | 1-15 minutes after spinal anesthesia
  The dose of prophylactic phenylephrine that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia.
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia.
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Base excess | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University